CLINICAL TRIAL: NCT03104049
Title: Pilot Study on the Effects of Neuromuscular Taping in Parkinson's Disease Patients
Acronym: NMT-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele Roma (Other)
Collaborators: Politecnico di Milano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RP 07/15
Record Dates: First submitted 2017-03-27; First posted 2017-04-07 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Neuromuscular taping; Trunk; Posture; Kinematic; rehabilitation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- the PD NMT Group (Active Comparator): the NMT Group were treated with NMT
  Interventions: Device: Neuromuscular taping
- The PD Group without NMT (No Intervention): The patients received only their usual pharmacological PD therapy

INTERVENTIONS:
Device: Neuromuscular taping — NMT applications:
  1. rhomboid major muscle
  2. muscles abdominals
  3. spinal muscles
  4. pectoralis major muscles
  5. gastrocnemius muscle
  6. upper trapezius muscle
  7. anterior muscles of the neck
  Other Names: NMT
  Arms: the PD NMT Group

SUMMARY:
Parkinson's disease (PD) is a degenerative disorder characterized by a symptom triad consisting on: tremor, rigidity and bradykinesia . To these symptoms it is often added postural alteration that can stand in two different attitudes, such as the camptocormia and the syndrome of Pisa . Progressing in its evolution, PD becomes increasingly disabling, making it difficult or even impossible daily activities such as washing or dressing.The abnormal posture, with alteration of the limbs, the neck and trunk, is a recurring feature in PD, with a frequency of about 30%. Between 2% and 12.3% are more severe abnormalities such as camptocormia, the syndrome of Pisa and the anterocollis. Several studies disease plug in Neuromuscular Taping technique (NMT) among rehabilitative tools in degenerative neurological syndromes.

To the best of our knowledge, no applications were found in PD. Therefore, the current study was designed to evaluate quantitatively the effects of the NMT intervention on the trunk kinematics during standing position. More specifically, this study aims to compare the trunk kinematic variables of patients with PD who were treated with effective NMT versus those of the subjects who received only the pharmacological treatment.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of idiopathic PD by United Kingdom Brain Bank criteria
* No other significant neurological or orthopedic problems
* Age between 55 and 80 years
* MDS-UPDRS item 3.13 Posture between mild and moderate (definite flexion, scoliosis or leaning to one side)
* Patient able to walk independently or with minimal assistance for 10 meters
* Medical treatment for Parkinson's Disease must be stable for at least two weeks prior to inclusion, and during the study. During the study, the dosage of anti-parkinsonian drug treatment should not change, if it is not deemed necessary by the investigator.

Exclusion criteria:

* Disability to understand instructions required by the study (Informed Consent Test of Comprehension)
* primarily wheelchair bound
* Skin abrasions
* sensitive skin

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 46 (Actual)
Dates: Start 2015-11-20 (Actual); Primary Completion 2016-12-18 (Actual); Study Completion 2017-01-08 (Actual)

PRIMARY OUTCOMES:
Change in the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) rating scale total score between baseline evaluations and end of treatment | baseline and end of treatment (1 month)
  Clinical measures were summarized as means and standard deviations for all the 46 patients.

SECONDARY OUTCOMES:
Change in the Parkinson Disease Quality of life 8 total score between baseline evaluations and end of treatment | baseline and end of treatment (1 month)
  Clinical measures were summarized as means and standard deviations for all the 46 patients.
Change in the Non Motor Symptoms scale total score between baseline evaluations and end of treatment | baseline and end of treatment (1 month)
  Clinical measures were summarized as means and standard deviations for all the 46 patients.
Change in the EuroQol 5 total score between baseline evaluations and end of treatment | baseline and end of treatment (1 month)
  Clinical measures were summarized as means and standard deviations for all the 46 patients.
Change in the Freezing of Gait total score between baseline evaluations and end of treatment | baseline and end of treatment (1 month)
  Clinical measures were summarized as means and standard deviations for all the 46 patients.

IPD SHARING:
Plan to Share IPD: Undecided